CLINICAL TRIAL: NCT02174211
Title: A Pharmacokinetic Study: Ranibizumab, Aflibercept and the Effect of Vitrectomy.
Acronym: VITCLEAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT Number: 2012-005500-18
Record Dates: First submitted 2014-06-24; First posted 2014-06-25 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A: Ranibizumab (Lucentis) (Active Comparator): Previous Vitrectomy
  Interventions: Drug: Ranibizumab
- Arm B: Ranibizumab (Lucentis) (Active Comparator): Non-vitrectomised, PVD / no PVD
  Interventions: Drug: Ranibizumab
- Arm C: Aflibercept (Eylea) (Active Comparator): Non-vitrectomised, PVD / no PVD
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal injection of ranibizumab
  Other Names: Lucentis
  Arms: Arm A: Ranibizumab (Lucentis); Arm B: Ranibizumab (Lucentis)
Drug: Aflibercept — Intravitreal injection of aflibercept
  Other Names: Eylea
  Arms: Arm C: Aflibercept (Eylea)

SUMMARY:
To study the effect of pars plana vitrectomy on the intravitreal pharmacokinetics of ranibizumab and to compare the half-life of ranibizumab and aflibercept.

DETAILED DESCRIPTION:
This study is a prospective, pharmacokinetic study comparing ranibizumab clearance in two groups of patients; those with and without prior vitrectomy. Additionally it will compare ranibizumab clearance to aflibercept clearance as well as the effect on systemic circulating inflammatory and safety markers. Patients will already be receiving ranibizumab or aflibercept therapy - the injection is itself administered irrespective of their participation in this study and therefore this study will not alter medical management or the choice of therapy.

To estimate ranibizumab and aflibercept clearance, it is important to measure serum concentrations at several intervals within the first 24 hours. Participants will ideally have venous blood sampling at the following times after their ranibizumab or aflibercept injection:

* 1 hour
* 2 hours
* 3 hours
* 4 hours
* 6 hours
* 24 hours
* 2 days
* 4 days
* 1 week*
* 2 weeks
* 4 weeks*

ELIGIBILITY:
Inclusion criteria

* Adults of either sex aged 55 years and older
* Active neovascular AMD in the study eye
* Intravitreal dose of 0.5 mg ranibizumab or 2 mg aflibercept required, as per current clinical guidelines
* Venous access that is sufficient to allow easy blood sampling on a frequent basis
* Able to give written consent
* Willingness to comply with all study procedures

Exclusion criteria

* Myopia greater than 8 dioptres in the study eye
* Axial length of eye under 20mm or over 26mm
* Aphakia in study eye
* Pseudophakia with a defect in the posterior capsule
* Glaucoma in study eye
* Current renal dialysis
* Presence of inflammatory eye conditions, such as uveitis, or systemic conditions likely to elevate CRP.
* Intraocular surgery within 6 months of enrolment, except for routine phacoemulsification cataract surgery that may occur within 4 months of enrolment
* Current treatment for wet age-related macular degeneration with an intravitreal agent other than ranibizumab or aflibercept in the study eye. Patients expected to change their anti-VEGF agent during the sampling period are also excluded.
* Known significant allergy to ranibizumab or aflibercept
* Participants who, in the opinion of the Investigator, would not be willing or able to comply with the study protocol or provide informed consent.
* Patients with severe anaemia
* Patients who have received anti-VEGF therapy in either eye within 8 weeks of enrolment, or who are likely to require anti-VEGF treatment in the fellow eye during the course of venous sampling. Note that the final venous sample at 4 weeks can be undertaken on the same day as an anti-VEGF injection, but must be taken prior to any injection.
* Patients presently taking any topical (skin or eye), periocular, intraocular, local or systemic treatment with immunosuppressive or anti-inflammatory agents, such as steroids, steroid sparing agents, and NSAIDs. Patients who have received any of these agents within 2 months prior to enrolment are also excluded, as are those thought likely to receive these medications during the course of venous sampling.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-06; Primary Completion 2020-11 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Ranibizumab half-life | 12 Months
  Vitrectomised and non-vitrectomised patients
Aflibercept half-life | 12 Months
  Non-vitrectomised patients only

SECONDARY OUTCOMES:
Sub-group analysis of the effect of PVD on ranibizumab half-life | 12 months
  Measurement of half-life (drug assay)
The effect of ranibizumab and aflibercept concentrations on serum inflammatory and safety marker levels. | 12 months
  Assay levels of cytokines and inflammatory/safety markers

CONTACTS AND LOCATIONS:
Overall Officials: Timothy L Jackson, PhD,FRCOphth, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital NHS Foundation Trust, London, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
The Investigator(s) shall permit trial-related monitoring, audits, REC review, and regulatory inspections (where appropriate) by providing direct access to source data and other documents (i.e. patients' case sheets, blood test reports, X-ray reports, histology reports etc). Where necessary, inspection may also take place at the site's facilities.